CLINICAL TRIAL: NCT05531435
Title: Local Anesthesia With SleeperOne® Device vs Traditional Syringe for Restorative Procedures in Pediatric Patients: Randomized Clinical Trial
Brief Title: Local Anesthesia With Computerized Device for Restorative Procedures in Pediatric Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pavia (Other)
Responsible Party: Principal Investigator, Andrea Scribante, Associate Professor, Principal Investigator, University of Pavia
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2022-SLEEPERONE
Record Dates: First submitted 2022-09-03; First posted 2022-09-08 (Actual); Last update posted 2022-09-22 (Actual); Status verified 2022-09

CONDITIONS: Dental Pain and Sensation Disorder; Dental Caries in Children
Keywords: dental anesthesia
MeSH Terms: conditions — Toothache; Sensation Disorders | interventions — Anesthesia, Local

STUDY DESIGN:
Intervention Model Description: Split-mouth design
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SleeperOne (Experimental): SleeperOne S4 (Revello S.p.A., Verona, Italy) appliance will be used for the administration of local anesthetic.
  Interventions: Drug: local anaesthetic injection
- Traditional anesthesia (Active Comparator): Local anesthesia will be performed with a traditional syringe (0480-1, ASA Dental, Massarosa, LU, Italy).
  Interventions: Drug: local anaesthetic injection

INTERVENTIONS:
Drug: local anaesthetic injection — Local anesthetic injection of articaine 4% + adrenaline 1/100.000 (Septanest, Septodont, Saint Maur des Fossés, France) with 30G - 9 mm needle (DENTAL HI TEC, ZI de l'Appentière, Mazières-en-Mauges, France).

SUMMARY:
The aim of the present study is to assess if there are differences on perceived pain during local anesthesia performed with SleeperOne device or with a traditional syringe in pediatric patients.

Patients responding to the inclusion criteria will be asked to participate to the study. After signing the informed consent, they will undergo local anesthesia procedure on first or second primary molars for the subsequent performing of dental filling. The split-mouth design will randomly allocate first or second primary molar from one quadrant to SleeperOne procedure, while the contralateral one will be subdued to local anesthesia with traditional syringe.

After the procedure, patients will be asked to assess the perceived pain with a Visual Analogue Scale from a range 0-10. VAS scales will be used to assess sensations of "size" (related to the two instruments), bitter and vomit.

DETAILED DESCRIPTION:
The aim of the present study is to assess if there are differences on perceived pain during local anesthesia performed with SleeperOne device or with a traditional syringe in pediatric patients.

Patients responding to the inclusion criteria will be asked to participate to the study. After signing the informed consent, they will undergo local anesthesia procedure on first or second primary molars for the subsequent performing of dental filling. Teeth will be randomly allocated to the two different local anesthesia types according to a split-mouth design: first or second primary molar from one quadrant will undergo SleeperOne anesthesia, while the contralateral one will undergo local anesthesia with traditional syringe.

After the procedure, patients will be asked to assess the perceived pain with a Visual Analogue Scale from a range 0-10. VAS scales will be used to assess sensations of size (related to the two instruments), bitter and vomit.

Sample size calculation (alfa = 0.05; power = 95%) for two independent study group and a continuous primary endpoint is performed concerning the primary outcome "VAS scale for pain". An expected mean of 2.6 with an expected mean difference of 1.7 and a standard deviation of 1.84 are hypothesized [Palm et al., 2004]; therefore, 30 teeth per group are required and a total of 30 patients for the split-mouth design study should be enrolled.

Statistical analysis will be performed. Data normality of distribution will be assessed with Kolmogorov-Smirnov test. Subsequently, the most appropriate test will be conducted to compare VAS differences between the two groups for the four variables "pain", "size", "bitter", "vomit".

Linear regressions will be performed to assess of the following independent variables on "pain", "size", "bitter" and vomit": technique, quadrant, dental arch, tooth, dentition, sex, age.

ELIGIBILITY:
Inclusion Criteria:

* presence of dental caries requiring filling with local anesthesia on first or second primary molar
* presence of dental caries requiring filling with local anesthesia on the contralateral primary molar

Exclusion Criteria:

* gingivitis
* dental abscesses, facial traumas/injuries
* drugs (NSAIDS, paracetamol, antibiotics)

Ages: 5 Years to 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 30 (Actual)
Dates: Start 2022-09-07 (Actual); Primary Completion 2022-09-21 (Actual); Study Completion 2022-09-21 (Actual)

PRIMARY OUTCOMES:
Pain measure | Baseline
  Self-reported pain by the patient immediately after local anesthesia infiltration using a VAS (visual analogue scale), containing a combination of Numeric Rating Scale (0-10, where 0 means no pain, 10 - worst possible pain) and Wong-Baker Faces Pain Scale, including pictures of facial expressions with correlating numbers of 0-10 (0 being 'no hurt' and 10 being 'hurts worst'). The combination allows children to pick a facial expression, that corresponds with their pain and see a number that matches it.

SECONDARY OUTCOMES:
Size sensation | Baseline
  Self-reported sensation of size related to the instruments by the patient after local anesthesia infiltration using a VAS (visual analogue scale), containing a combination of Numeric Rating Scale (0-10, where 0 means no size, 10 - very bulky) and Wong-Baker Faces Pain Scale, including pictures of facial expressions with correlating numbers of 0-10 (0 being 'no problem with it' and 10 being 'very bulky'). The combination allows children to pick a facial expression, that corresponds with their sensation and see a number that matches it.
Bitter sensation | Baseline
  Self-reported sensation of bitter by the patient after local anesthesia infiltration using a VAS (visual analogue scale), containing a combination of Numeric Rating Scale (0-10, where 0 means no bitter, 10 - very bitter) and Wong-Baker Faces Pain Scale, including pictures of facial expressions with correlating numbers of 0-10 (0 being 'no bitter' and 10 being 'very bitter'). The combination allows children to pick a facial expression, that corresponds with their sensation and see a number that matches it.
Vomit sensation | Baseline
  Self-reported sensation of vomit by the patient after local anesthesia infiltration using a VAS (visual analogue scale), containing a combination of Numeric Rating Scale (0-10, where 0 means no vomit, 10 - very vomiting at all) and Wong-Baker Faces Pain Scale, including pictures of facial expressions with correlating numbers of 0-10 (0 being 'no vomit' and 10 being 'very vomiting'). The combination allows children to pick a facial expression, that corresponds with their sensation and see a number that matches it.

CONTACTS AND LOCATIONS:
Overall Officials: Andrea Scribante, DDS, PhD, Principal Investigator — University of Pavia
Locations (1):
- Unit of Orthodontics and Pediatric Dentistry - Section of Dentistry - Department of Clinical, Surgical, Diagnostic and Pediatrics - University of Pavia, Pavia, Lombardy, Italy

IPD SHARING:
Plan to Share IPD: No
Data will be available upon motivated request to the Principal Investigator.

REFERENCES:
- [Background] Palm AM, Kirkegaard U, Poulsen S. The wand versus traditional injection for mandibular nerve block in children and adolescents: perceived pain and time of onset. Pediatr Dent. 2004 Nov-Dec;26(6):481-4. PMID 15646908